CLINICAL TRIAL: NCT05301725
Title: Efficacy of Different Acid Suppressors in Bismuth-containing Quadruple Therapy as First-line Treatment Against Helicobacter Pylori
Brief Title: Efficacy of Different Acid Suppressors in Bismuth-containing Quadruple Therapy Against Helicobacter Pylori
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of Qilu Hospital gastroenterology department, Shandong University
Other Study IDs: 2022-SDU-QILU-G001
Record Dates: First submitted 2022-02-14; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Helicobacter Pylori; Eradication Rate
Keywords: Helicobacter pylori,eradication therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PPI group: PPI regimen
  Interventions: Other: PPI regimen
- P-CAB group: P-CAB regimen
  Interventions: Other: P-CAB regimen

INTERVENTIONS:
Other: PPI regimen — All patients received PPI regimen( lansoprazole or esomeprazole,bismuth amoxicillin,clarithromycin for14 days). Demographic data,treatment regimens, outcomes of therapy, adherence to therapy and adverse event were retrieved.
  Groups: PPI group
Other: P-CAB regimen — All patients received P-CAB regimen(vonoprazan,bismuth ,amoxicillin,clarithromycin for14 days). Demographic data,treatment regimens, outcomes of therapy, adherence to therapy and adverse event were retrieved.
  Groups: P-CAB group

SUMMARY:
Ａretrospective study was conducted to compare the efficacy, safety, and cost-effectiveness of traditional proton pump inhibitors (PPI ) and Potassium-competitive acid blockers ( P-CAB )for clarithromycin-based bismuth-containing quadruple therapy in the management of Helicobacter pylori eradication.

DETAILED DESCRIPTION:
This study retrospectively enrolled participants with H. pylori infection who received bismuth quadruple regimen containing clarithromycin. The basic information, treatment results, adverse reactions and compliance of the patients were collected. According to the type of acid inhibitors, participants were divided into traditional PPI group and P-CAB group. Traditional PPI group which were divided into lansoprazole group and esomeprazole group. The eradication rate, safety, compliance of H. pylori in different treatment regimens was evaluated. Multivariate analysis was performed to identify predictors of eradication failure.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-75 years with persistent H. pylori infection.
* Participants received clarithromycin-based bismuth-containing quadruple therapy.

Exclusion Criteria:

* Patients received rescue therapy
* Patients treated with PPI, P-CAB,bismuth and antibiotics in the previous 4 weeks
* Patients with gastorectomy
* Currently pregnant or lactating or other conditions unable to receive therapy
* Severe concomitant cardiovascular, respiratory, or endocrine diseases, clinically significant renal or hepatic disease, hematologic disorders and any other clinically significant medical condition that could increase risk
* Severe neurologic or psychiatric disorders
* Information incomplete

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: helicobacter infection
Sampling Method: Non-Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of eradication success | 1 month
  Six weeks after completion of treatment, numbers of patients get H.pylori eradicated supported by negative 13C-UBT results will be investigated by an independent researcher. Then eradication rate in each group will be calculated by using intention-to-treat (ITT) analysis, modified intention to treat analysis (MITT) and per-protocol (PP) analysis. The ITT analysis includes all the patients who take at least one dose of the study medications. The MITT analysis is limited to patients who complete follow-up.The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.
Prevalence of adverse events | 1 month
  At the follow-up, adverse events complained by patients will be recorded by an independent researcher, meanwhile CTCAE v5.0 was used to evaluate severity of adverse events.The prevalence of adverse events was compared between the two group
Number of participants with good compliance | 1 month
  Compliance was evaluated by assessing the total pills patients have taken.Compliance was defined as good whenmore than 90% or less than 120% of the total pills were taken

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hosipital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang J, Li YY, Lin MJ, Liu J, Lin BS, Ding YM, Wan M, Zhang WL, Kong QZ, Wang ST, Mu YJ, Duan M, Han ZX, Zuo XL, Li YQ. Vonoprazan is noninferior to proton pump inhibitors in bismuth-containing quadruple therapy for the treatment of Helicobacter pylori infection: A propensity score matching analysis. J Dig Dis. 2023 Jan;24(1):19-27. doi: 10.1111/1751-2980.13166. Epub 2023 Apr 22. PMID 36960538